CLINICAL TRIAL: NCT00366223
Title: Changing Patterns of Candida Infections in Urban Medical Centers: Emphasis on the Emergence of Non-albicans Species and Their Influence on Clinical Outcomes
Brief Title: Changing Patterns of Candida Infections in Urban Medical Centers
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB#0607092
Record Dates: First submitted 2006-08-18; First posted 2006-08-21 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Infection; Candida; Non Albicans Species
Keywords: infection; candida
MeSH Terms: conditions — Infections; Torulopsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — No genetic testing will be performed on any of the samples being obtained. The biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed. All samples will be kept in the investigator's laboratory located in Scaife Hall, Room 812, 3550 Terrace Street.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the changing patterns of infection caused by Candida species in urban medical centers and its influence on patient outcomes. A retrospective cohort study design will be employed with the main outcome measure being hospital mortality. Secondary outcomes including microbiologic clearance of the infection, duration of hospitalization, and the intensive care unit (ICU) length of stay will also be assessed.

DETAILED DESCRIPTION:
The following information that was collected as part of the patient's clinical treatment will be collected: age, sex, occupation, hospital location at the time of positive culture (ER, medical ward, ICU, etc.), prior hospitalization, receipt of outpatient dialysis, home care or other regular medical care (eg, outpatient chemotherapy), presence of invasive devices, receipt of antibiotics, including their type and whether they were adequate for the resistance profile of the organism, prior positive microbiologic cultures, time and location of positive cultures, underlying diseases and severity of illness, presence of urinary or intravascular devices, recent immunomodulative therapies or radiation therapy, physical exam findings, laboratory and radiographical data, antimicrobial usage within 30 days of onset of the infection, microbiological data and resistance patterns, choice of antibiotics once organism identified, bacteriological outcomes, laboratory results, demographic information, medications, clinical outcome, gender, height, weight, ethnicity, and past medical history. We will collect information retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* All hospitalized patients with a positive blood culture for Candida will be eligible.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: candida blood culture
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
dead or alive | end of study
  Health status

CONTACTS AND LOCATIONS:
Overall Officials: David L Paterson, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States